CLINICAL TRIAL: NCT07296614
Title: Integrative Chinese and Western Medicine for Diminished Ovarian Reserve-Associated Infertility in Natural Conception Population
Brief Title: Clinical Evaluation of Integrated Chinese-Western Medicine for Infertility With DOR Patients in Women Achieving Natural Pregnancy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Dongfang Hospital Beijing University of Chinese Medicine (Other); Beijing University of Chinese Medicine (Other); The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Hunan University of Traditional Chinese Medicine (Other); Shandong University (Other); Xiamen University (Other); Beijing Obstetrics and Gynecology Hospital (Other); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); The Third Affiliated Hospital of Beijing University of Chinese Medicine (Other); Hunan Provincial Maternal and Child Health Care Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); The Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Unknown); Institute of Basic Medical Sciences CAMS (Unknown); First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); Shunde Women and Children's Hospital (Maternity and Child Healthcare Hospital of Shunde Foshan) (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Shenyang Women's and Children's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K9220
Record Dates: First submitted 2025-11-28; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Diminished Ovarian Reserve (DOR); Infertility
Keywords: Diminished ovarian reserve (DOR); Infertility; Integrated Traditional Chinese and Western Clinical Medicine; Randomized controlled trial
MeSH Terms: conditions — Infertility | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Western medicine group (Placebo Comparator): Take the placebo granules orally for three months, followed by three cycles of letrozole while continuing the placebo.
  Interventions: Drug: Western Medicine; Drug: Placebo
- Integrated traditional Chinese and Western medicine (Experimental): Take the "Xiehe DOR Kidney-Tonifying Universal Formula" orally for three months; thereafter, continue the Chinese herbal formula while combining it with three cycles of letrozole.
  Interventions: Drug: Western Medicine; Drug: Traditional Chinese Medicine

INTERVENTIONS:
Drug: Western Medicine — Letrozole is administered orally at 2.5 mg once daily from Day 2 to Day 5 of the menstrual cycle (5 consecutive days).
Drug: Traditional Chinese Medicine — "Xiehe DOR Kidney-Tonifying Universal Formula" is a traditional Chinese medicine (TCM) granule formulation prepared in-hospital. It is taken by dissolving one sachet in hot water, three times daily.
  Arms: Integrated traditional Chinese and Western medicine
Drug: Placebo — The appearance and packaging of the placebo are exactly the same as those of "Xiehe DOR Kidney-Tonifying Universal Formula". It is also taken by dissolving one sachet in hot water, three times daily.
  Arms: Western medicine group

SUMMARY:
This study aims to evaluate the superiority of an integrated traditional Chinese and Western medicine regimen ("Xiehe DOR Bushen Tongzhi Formula" + ovulation induction therapy with ovulation monitoring and timed intercourse) compared to standard treatment alone (placebo + ovulation induction therapy with ovulation monitoring and timed intercourse) in improving the natural cumulative clinical pregnancy rate in infertile patients with kidney deficiency-type diminished ovarian reserve (DOR).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 22 to 39 years (inclusive).
2. Meet the diagnostic criteria for diminished ovarian reserve (requiring at least two of the following: Basal FSH 10-25 IU/L; AMH < 1.1 ng/mL; AFC < 7) and infertility(defined as the failure to achieve pregnancy after 12 months of regular unprotected sexual intercourse).
3. Meet the diagnostic criteria for kidney deficiency syndrome in traditional Chinese medicine
4. Voluntarily participate in this study and provide written informed consent.

Exclusion Criteria:

1. Patients with premature ovarian insufficiency or premature ovarian failure (basal FSH >25 IU/L), organic pathologies such as ovarian tumors, endometrial tuberculosis, intrauterine adhesions, or endometrial injuries, as well as those with congenital adrenal hyperplasia or Cushing's syndrome;
2. Infertility caused by organic lesions of the fallopian tubes, uterus, cervix, etc.
3. Infertility due to male factors (based on semen analysis reports, meeting the diagnostic criteria for oligoasthenoteratozoospermia according to the WHO 5th edition standards).
4. DOR caused by iatrogenic factors (such as pelvic surgery, radiotherapy/chemotherapy, uterine artery embolization, etc.).
5. Patients with severe primary diseases of the cardiovascular, cerebrovascular, hepatic, renal, or hematopoietic systems, or psychiatric disorders.
6. Individuals with known allergies to the investigational drug or its components.
7. Use of hormonal medications (e.g., estrogen, contraceptive drugs) within one month prior to enrollment, or use of kidney-tonifying Chinese herbal medicines or proprietary Chinese medicinal products within one month prior to enrollment.
8. Patients currently participating in or planning to participate in other clinical trials.

Ages: 22 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative clinical pregnancy rate | Assessed at study completion, approximately 6 months after enrollment.
  The rate of intrauterine pregnancy confirmed by transvaginal ultrasound

SECONDARY OUTCOMES:
Indicators related to ovarian reserve function | Baseline, 3-months, 6-months
  sex hormone levels(AMH, FSH), antral follicle count(AFC)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No